CLINICAL TRIAL: NCT04170023
Title: A Phase 2 Open-Label Proof of Concept Study to Assess the Efficacy, Safety, and Pharmacokinetics of the Oral Factor D (FD) Inhibitor ALXN2050 (ACH-0145228) in Paroxysmal Nocturnal Hemoglobinuria (PNH) Patients as Monotherapy
Brief Title: Study of the Oral Factor D (FD) Inhibitor ALXN2050 in PNH Patients as Monotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not appropriately control IVH; significantly increased rates of BTH and LDH excursions (LDH excursions is defined by LDH values > X2ULN) compared to ravulizumab.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACH228-110; 2019-003830-17 (EudraCT Number)
Record Dates: First submitted 2019-11-06; First posted 2019-11-20 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: paroxysmal nocturnal hemoglobinuria; PNH; extravascular hemolysis; EVH; factor D inhibitor; complement; C5 inhibitor; danicopan
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Hemolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label ALXN2050 Monotherapy (Experimental): Experimental: Open-label ALXN2050 Monotherapy ALXN2050 orally administered
  Group 1: Patients with PNH who are treatment naïve
  Group 2: Patient with PNH who have received complement component 5 (C5) inhibition with eculizumab for at least 6 months, who continue to experience anemia and reticulocytes above the upper limit of normal (ULN)
  Group 3: Patients with PNH who have received danicopan monotherapy during study ACH471-103
  Interventions: Drug: ALXN2050

INTERVENTIONS:
Drug: ALXN2050 — Oral FD inhibitor
  Other Names: ACH-0145228

SUMMARY:
The study will evaluate the efficacy and safety of the oral Factor D (FD) inhibitor ALXN2050 (ACH-0145228) monotherapy in patients with PNH that are treatment naïve, or patients currently treated with eculizumab who still experience anemia and reticulocytosis, or patients currently treated with ALXN2040 (danicopan) as monotherapy. After signing consent, participants will have periodic visits through Week 12, at which time the primary endpoint and key secondary assessments will be analyzed. Participants will continue on treatment past 12 weeks into a long-term extension portion of the trial.

DETAILED DESCRIPTION:
Experimental: Open-label ALXN2050 Monotherapy orally

Group 1: Patients with PNH who are treatment naïve

Group 2: Patients with PNH who have received complement component 5 (C5) inhibition with eculizumab for at least 6 months, who continue to experience anemia and reticulocytes above the upper limit of normal (ULN) who will switch to ALXN2050 monotherapy

Group 3: Patients with PNH receiving danicopan monotherapy in study ACH471-103 will switch to ALXN2050 monotherapy

After signing the informed consent form, participants will enter the screening period. During the Screening Period, eligibility and screening assessments will be performed. Screening assessments may be spread over more than one visit if necessary. At the baseline visit, screened participants who continue to meet eligibility criteria will enter the Treatment Period.

The treatment phase will be followed by a long-term extension phase, where ALXN2050 will continue to be administered.

Blood will be collected to assess the efficacy endpoints, such as, change in hemoglobin (Hgb), lactate dehydrogenase (LDH), and other measures of hemolysis. Safety and transfusion requirements will also be assessed.

Participants will continue on treatment past 12 weeks in a long-term extension portion of the trial.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of PNH.
2. Male or female, ≥ 18 years of age

Eligibility Criteria:

Eligibility Criteria Specific for Group 1:

1. PNH Patients who have no history of treatment with any complement inhibitor at any dose.
2. PNH Type III erythrocyte or granulocyte clone size ≥10%
3. Absolute reticulocyte count ≥100×10^9/liter [L].
4. Anemia (Hgb <10.5 grams/deciliter [g/dL]).
5. LDH ≥1.5× upper limit of normal.
6. Platelet count ≥30,000/microliter (µL)
7. Absolute neutrophil count (ANC) ≥750/ µL.

Eligibility Criteria Specific for Group 2:

1. Stable background regimen of at least 24 weeks for eculizumab without change in dose or interval for at least the past 8 weeks
2. Anemia (Hgb <10 g/dL)
3. Absolute reticulocyte count ≥100×10^9/L
4. Platelet count ≥30,000/µL
5. Absolute neurophil count (ANC) ≥750/ µL

Eligibility Criteria Specific for Group 3:

1. Patient received danicopan during Study ACH471-103

Key Exclusion Criteria:

1. History of a major organ transplant or hematopoietic stem cell/marrow transplant .
2. Known aplastic anemia or other bone marrow failure that requires HSCT, or if these patients are on immunosuppressive agents for less than 24 weeks.
3. Known underlying bleeding disorders or any other conditions leading to anemia not primarily associated with PNH.
4. Estimated glomerular filtration rate <30 milliliters/minute/1.73 meters squared and/or are on dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2024-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Lévis, Quebec
- Italy (2):
  - Research Site, Avellino
  - Research Site, Florence
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Grafton
- Research Site, Seoul, South Korea
- Research Site, Albacete, Spain
- Turkey (Türkiye) (2):
  - Research Site, Istanbul
  - Research Site, Izmir
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Kulasekararaj AG, Browett PJ, Risitano AM, Patriquin CJ, Yenerel MN, Marceau D, Sahin F, Algarra L, Ogawa M, Yu J, Cross N, Notaro R, Lee JW, Brodsky RA. Efficacy and Safety of Vemircopan as Monotherapy in Patients With Paroxysmal Nocturnal Hemoglobinuria. Blood Adv. 2025 Oct 22:bloodadvances.2025017731. doi: 10.1182/bloodadvances.2025017731. Online ahead of print. PMID 41124654
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACH228-110&attachmentIdentifier=b24b7f34-0fe7-4d98-b59a-1802bfcdd0ed&fileName=ACH228-110_CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a 12-week Treatment Period and a 148-week or 200-week (for sites in New Zealand) Long-term Extension (LTE) Period.
Groups:
- Group 1: Treatment Naive: Participants who were treatment-naive received ALXN2050 orally for 12 weeks during the treatment period. At the end of Week 12, participants entered the 148-week LTE Period and continued to receive ALXN2050 orally.
- Group 2: Eculizumab Switch: Participants who had received component 5 (C5) inhibition with eculizumab for at least 6 months, who continued to experience anemia (hemoglobin [Hgb] <10 grams/deciliter [dL]) and reticulocytes above the upper limit of normal (ULN), switched to ALXN2050 in this study and received ALXN2050 orally for 12 weeks during the treatment period. At the end of Week 12, participants entered the 148-week LTE Period and continued to receive ALXN2050 orally.
- Group 3: Danicopan Rollover: Participants who had received danicopan monotherapy during Study ACH471-103 (NCT03181633), switched to ALXN2050 in this study and received ALXN2050 orally for 12 weeks during the treatment period. At the end of Week 12, participants entered the 148-week LTE Period and continued to receive ALXN2050 orally.
Period: Treatment Period
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Started | 12 | 11 | 6
Received at Least 1 Dose of Study Drug | 12 | 11 | 6
Completed | 12 | 11 | 6
Not Completed | 0 | 0 | 0
Period: LTE Period
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Started | 12 | 11 | 6
Received at Least 1 Dose of Study Drug | 12 | 11 | 6
Completed | 0 | 0 | 1
Not Completed | 12 | 11 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Study Termination | 11 | 11 | 5

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 dose of ALXN2050 in this study.
Groups:
- Group 2: Eculizumab Switch: Participants who had received C5 inhibition with eculizumab for at least 6 months, who continued to experience anemia (Hgb <10 grams/dL) and reticulocytes above the ULN, switched to ALXN2050 in this study and received ALXN2050 orally for 12 weeks during the treatment period. At the end of Week 12, participants entered the 148-week LTE Period and continued to receive ALXN2050 orally.
- Total: Total of all reporting groups
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover | Total
Number analyzed (Participants) | 12 | 11 | 6 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.75 (17.099) | 42.45 (13.419) | 40.50 (16.718) | 42.59 (15.186)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 3 | 14
  Male | 8 | 4 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 10 | 6 | 28
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 8 | 1 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 10 | 6 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
HgB [Mean (Standard Deviation); unit: grams/liter] | 81.17 (11.731) | 91.00 (9.602) | 130.67 (19.180) | 95.14 (22.662)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hgb at Week 12
Description: Hgb baseline was defined as the lowest Hgb value observed between and including screening and first dose date. To address the impact of transfusion, Hgb values collected within 4 weeks after transfusion were not included in the primary efficacy analysis. Change from Baseline = Hgb at Week 12 - Baseline Hgb.
Time Frame: Baseline, Week 12
Population: Full analysis set included all participants who received at least 1 dose of ALXN2050 in this study. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: grams/liter
Groups:
- Group 1: Treatment Naive: Participants who were treatment-naive received ALXN2050 orally for 12 weeks during the treatment period.
- Group 2: Eculizumab Switch: Participants who had received C5 inhibition with eculizumab for at least 6 months, who continued to experience anemia (Hgb <10 grams/dL) and reticulocytes above the ULN, switched to ALXN2050 in this study and received ALXN2050 orally for 12 weeks during the treatment period.
- Group 3: Danicopan Rollover: Participants who had received danicopan monotherapy during Study ACH471-103 (NCT03181633), switched to ALXN2050 in this study and received ALXN2050 orally for 12 weeks during the treatment period.
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 11 | 10 | 6
grams/liter | 35.6 (14.70) | 32.5 (20.03) | -3.7 (15.77)

2. Secondary Outcome: Number of Participants Who Had Transfusion Avoidance During 12 Weeks of Treatment With ALXN2050
Description: Transfusion avoidance: participants remained transfusion-free and did not require a transfusion during the period of interest.
Time Frame: Baseline up to Week 12
Population: Full analysis set included all participants who received at least 1 dose of ALXN2050 in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 12 | 11 | 6
Participants | 9 | 10 | 5

3. Secondary Outcome: Number of Red Blood Cell (RBC) Units Transfused During 12 Weeks of Treatment
Time Frame: Baseline up to Week 12
Population: Full analysis set included all participants who received at least 1 dose of ALXN2050 in this study.
Measure: Mean (Standard Deviation); unit: RBC units
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 12 | 11 | 6
RBC units | 0.6 (1.24) | 0.1 (0.30) | 0.8 (2.04)

4. Secondary Outcome: Number of Transfusion Instances During 12 Weeks of Treatment
Time Frame: Baseline up to Week 12
Population: Full analysis set included all participants who received at least 1 dose of ALXN2050 in this study.
Measure: Mean (Standard Deviation); unit: transfusion instances
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 12 | 11 | 6
transfusion instances | 0.4 (0.90) | 0.1 (0.30) | 0.5 (1.22)

5. Secondary Outcome: Change From Baseline in Lactate Dehydrogenase (LDH) at Week 12
Description: Change from Baseline = Serum LDH levels at Week 12 - Baseline Serum LDH levels.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 11 | 11 | 6
units/liter | -1310.8 (424.89) | 160.2 (279.57) | 88.7 (265.00)

6. Secondary Outcome: Change From Baseline in Absolute Reticulocyte Count at Week 12
Description: Change from Baseline = absolute reticulocyte count at Week 12 - Baseline reticulocyte count.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter (μL)
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 12 | 10 | 5
10^3 cells/microliter (μL) | -100.6 (72.18) | -179.0 (117.30) | -24.0 (22.10)

7. Secondary Outcome: Change From Baseline in Direct and Total Bilirubin at Week 12
Time Frame: Baseline, Week 12
Population: Full analysis set included all participants who received at least 1 dose of ALXN2050 in this study. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: micromoles (μmol)/liter
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 11 | 11 | 6
micromoles (μmol)/liter
  Direct Bilirubin: number analyzed (Participants) | 8 | 11 | 5
  Direct Bilirubin | -2.1 (2.10) | -6.3 (5.16) | 0.4 (0.89)
  Total Bilirubin | -12.9 (10.07) | -23.3 (24.89) | 1.5 (2.81)

8. Secondary Outcome: Change From Baseline in Paroxysmal Nocturnal Hemoglobinuria (PNH) Red Blood Cell (RBC) Clone Size at Week 12
Description: The PNH RBC clone size refers to the percentage of PNH-affected cells versus normal cells within the total cell population. Change from Baseline = PNH clone size at Week 12 - Baseline PNH clone size.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of the total cell population
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 9 | 3 | 2
percentage of the total cell population | 41.9 (13.68) | 27.5 (21.60) | -12.0 (26.94)

9. Secondary Outcome: Change From Baseline in Component 3 (C3) Fragment Deposition on PNH RBCs at Week 12
Description: C3 fragment deposition on PNH RBC was used as a marker of intra and extravascular hemolysis. Data are presented for the change from baseline to Week 12 in percentage of PNH RBCs with C3 fragment deposition.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of PNH RBC
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 10 | 3 | 2
percentage of PNH RBC | 0.0 (0.00) | -388.6 (590.08) | 0.3 (0.35)

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Events Leading to Discontinuation of Study Medication
Description: An adverse event (AE) was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), or an important medical event or reaction. A TEAE was defined as an AE that emerged during treatment, had been absent prior to treatment, or worsened relative to the pretreatment state. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: From first dose of study drug up to Week 217
Population: Safety set included all participants who received at least 1 dose of ALXN2050 in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 12 | 11 | 6
Participants
  Any AEs | 12 | 10 | 6
  SAEs | 7 | 5 | 2
  AEs Leading to Discontinuation of Study Medication | 1 | 1 | 0

11. Secondary Outcome: Change From Baseline in Hgb at the End of Treatment (EOT) During the LTE Period
Description: Hgb baseline was defined as the lowest Hgb value observed between and including screening and first dose date. Change from Baseline = Hgb at the EOT visit - Baseline Hgb.
Time Frame: Baseline, EOT visit (Maximum exposure: 213.4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams/liter
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 10 | 8 | 5
grams/liter | 44.9 (21.07) | 32.5 (7.17) | 2.4 (19.44)

12. Secondary Outcome: Change From Baseline in LDH at the EOT During the LTE Period
Description: Change from Baseline = Serum LDH levels at the EOT visit - Baseline Serum LDH levels.
Time Frame: Baseline, EOT visit (Maximum exposure: 213.4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units/liter
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 11 | 10 | 5
units/liter | -1084.1 (738.26) | 95.7 (223.88) | -61.4 (62.85)

13. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale (Version 4) Total Score at Week 12
Description: The FACIT-Fatigue scale is a collection of quality-of-life questionnaires pertaining to the management of fatigue symptoms due to chronic illness. The FACIT-Fatigue is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the preceding 7 days. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). Total scores ranged from 0 to 52, with higher score indicating better quality of life.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 11 | 7 | 6
units on a scale | 11.2 (13.20) | 5.1 (8.47) | 0.2 (3.13)

14. Secondary Outcome: Change From Baseline in FACIT-Fatigue Scale (Version 4) Total Score at the EOT During the LTE Period
Description: as for outcome 13
Time Frame: Baseline, EOT visit (Maximum exposure: 213.4 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
Number analyzed (Participants) | 11 | 9 | 5
units on a scale | 12.6 (12.51) | 4.4 (7.26) | -3.4 (10.26)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 217
Description: Safety set included all participants who received at least 1 dose of ALXN2050 in this study.
Arm/Group | Group 1: Treatment Naive | Group 2: Eculizumab Switch | Group 3: Danicopan Rollover
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/6
Serious Adverse Events (participants affected / at risk) | 7/12 | 5/11 | 2/6
Other Adverse Events (participants affected / at risk) | 12/12 | 10/11 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Treatment Naive (N=12) | Group 2: Eculizumab Switch (N=11) | Group 3: Danicopan Rollover (N=6)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 4 | 2 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0
Haemoglobinuria (Renal and urinary disorders) | 1 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Intravascular haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Treatment Naive (N=12) | Group 2: Eculizumab Switch (N=11) | Group 3: Danicopan Rollover (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Breakthrough haemolysis (Blood and lymphatic system disorders) | 3 | 2 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 4 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Episcleritis (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Tongue geographic (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2 | 0
Catheter site rash (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 2 | 0
Fatigue (General disorders) | 6 | 1 | 3
Influenza like illness (General disorders) | 1 | 2 | 2
Vaccination site pain (General disorders) | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 2 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 2 | 0
Pulpitis dental (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood creatine increased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 3 | 1
International normalised ratio increased (Investigations) | 0 | 1 | 0
Liver function test increased (Investigations) | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 2
Headache (Nervous system disorders) | 6 | 3 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 2 | 1 | 2
Haematuria (Renal and urinary disorders) | 3 | 4 | 2
Haemoglobinuria (Renal and urinary disorders) | 3 | 2 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Intravascular haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1
Exudative retinopathy (Eye disorders) | 1 | 0 | 0
Retinal degeneration (Eye disorders) | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Hyperthermia (General disorders) | 2 | 0 | 0
Malaise (General disorders) | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 2 | 2
Rebound effect (General disorders) | 1 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 4 | 2 | 3
Cellulitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Furuncle (Infections and infestations) | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0 | 0
Tinea versicolour (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0
Epstein-Barr virus antibody positive (Investigations) | 0 | 1 | 0
Free haemoglobin present (Investigations) | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 2 | 1 | 0
Low density lipoprotein increased (Investigations) | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 0 | 0
Sleep disorder (Psychiatric disorders) | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Choluria (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT04170023/Prot_002.pdf
  • Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT04170023/SAP_001.pdf